CLINICAL TRIAL: NCT07150468
Title: Establishment of a Strategy for Preventing Graft-versus-host Disease After Allogeneic Hematopoietic Cell Transplantation by Exploring Immune Mechanisms of Regulatory and Effector T Cells
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yunsuk Choi, Associate professor, Asan Medical Center
Other Study IDs: preventing GVHD after allo-HCT
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Leukemia, Myelodysplastic Syndrome, Myeloproliferative Neoplasms, Lymphoma, Multiple Myeloma
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma; Multiple Myeloma | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sampling blood — Sampling
  1. patient
     1. Peripheral blood samples in a volume of 25 cc will be collected before HCT and 2 weeks after HCT, and peripheral blood samples in a volume of 20 cc will be collected 4 weeks, 3 months, 6 months, and 12 months after HCT.
     2. If GVHD occurs, additional blood sample (20 cc) will be collected.
     3. In case of organ-specific GVHD including skin, gut, liver, muscle, etc., tissue samples from biopsy will be obtained for further analysis.
  2. donor a. Peripheral blood samples in a volume of 20 cc will be collected before HCT

SUMMARY:
The purpose of this study was to explore the regulatory and effector T cell-related immune mechanisms associated with the development of graft-versus-host disease (GVHD) after allogeneic hematopoietic cell transplantation (HCT) using patient-derived derivatives, thereby establishing the basis for GVHD prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients: Patients aged 16 to 75 years receiving allogeneic hematopoietic stem cell transplantation for hematologic malignancies at Seoul Asan Medical Center.

2. Family members: Family members of patients under 75 years of age who meet Criterion 1 and are willing to donate peripheral blood hematopoietic stem cells.

Exclusion Criteria:

* Patients receiving cord blood transplantation.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients and family donors undergoing allogeneic hematopoietic cell transplantation at Seoul Asan Medical Center
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Immune cell phenotype analysis | before HCT and 2 weeks after HCT, 4 weeks, 3 months, 6 months, and 12 months after HCT. If GVHD occurs
  Immune cell phenotypes will be analyzed by examining immunophenotypic changes in regulatory T cells and acquired immune cells using a 6-color flow cytometer. For skin and intestinal graft-versus-host disease tissues, multi-color imaging techniques (e.g., Polaris, CODEX) will be utilized to obtain spatial information and the pathogenic potential of various immune cells within the tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided